CLINICAL TRIAL: NCT02451566
Title: TriVascular Canadian LIFE Study: Least Invasive Fast-Track EVAR With the Ovation Prime™ Abdominal Stent Graft System
Brief Title: TriVascular Canadian LIFE Study: Least Invasive Fast-Track EVAR (Endovascular Aneurysm Repair)
Status: Completed | Type: Observational
Sponsor: TriVascular, Inc. (Industry)
Responsible Party: Sponsor
Organization: Endologix (Industry)
Other Study IDs: 771-0017
Record Dates: First submitted 2015-05-18; First posted 2015-05-22 (Estimated); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal; Aortic; Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Fast-Track Group: Includes subject who complete the Fast-Track EVAR protocol.
  Interventions: Device: Ovation Prime Abdominal Stent Graft System
- Standard P-EVAR Group: Includes subjects who do not complete the Fast-Track EVAR protocol, and their procedures are completed with bilateral percutaneous access.
  Interventions: Device: Ovation Prime Abdominal Stent Graft System
- Standard EVAR Group: Includes subjects who do not complete the Fast-Track EVAR protocol, and their procedures are not completed with bilateral percutaneous access (i.e. converted to femoral cutdown or open surgical repair).
  Interventions: Device: Ovation Prime Abdominal Stent Graft System

INTERVENTIONS:
Device: Ovation Prime Abdominal Stent Graft System

SUMMARY:
The primary objectives of the LIFE Study are to demonstrate the clinical cost and benefits associated with using the Ovation Prime Abdominal Stent Graft System under the least invasive conditions defined in the Fast-Track EVAR protocol. The key elements of the Fast-Track EVAR protocol include: appropriate patient selection, bilateral percutaneous access, no general anesthesia, no ICU admission post procedure, and next day discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years of age.
2. Patients who are male or non-pregnant female (females of child bearing potential must have a negative pregnancy test prior to enrollment into the study).
3. Patient has signed a Research Ethics Board (REB) approved Informed Consent Form.
4. Patient is considered by the treating physician to be a candidate for elective open surgical repair of the AAA (i.e., category I, II, or III per American Society of Anesthesiology (ASA) classification; refer to Appendix III: ASA Classification System).
5. Patient has an infrarenal abdominal aortic aneurysm that meets at least one of the following:

   * Abdominal aortic aneurysm >5cm in diameter
   * Aneurysm has increased in size by 0.5cm in last 6 months
   * Maximum diameter of aneurysm exceeds 1.5 times the transverse dimension of an adjacent non-aneurysmal aortic segment
6. Patient has suitable anatomy that allows use of the TriVascular Ovation/Ovation Prime Abdominal Stent Graft System:

   * Iliac or femoral arteries that allow endovascular access with the TriVascular Ovation/Ovation Prime Abdominal Stent Graft System (14F OD).
   * Proximal aortic neck landing zone with an inner wall diameter of no less than 16 mm and no greater than 30 mm at 13 mm below the inferior renal artery.
   * Proximal aortic neck with a length of at least 7 mm proximal to the aneurysm
   * Distal iliac artery landing zone an inner wall diameter of no less than 8 mm and no greater than 20 mm.
   * Distal iliac artery landing zone an inner wall diameter of no less than 8 mm and no greater than 20 mm.
   * Distance from the most distal renal artery to most superior internal iliac artery measurement is at least 130 mm.
7. Patient has suitable femoral arteries at the percutaneous access site that allow use of the Perclose ProGlide Suture-Mediated Closure (SMC) System via the pre-close technique, including:

   * ≥5 mm in diameter
   * At least 2 cm segment for access, 10 mm above the origin of the profunda femoris branch and 10 mm below the lower margin of the inferior epigastric artery as determined on preoperative contrast-enhanced CT, angiography, or ultrasound.
   * No calcification on the anterior wall or circumferential (>50%) calcification on the posterior wall.
   * No prior groin incision, hematoma, or significant scarring.
   * No prior clip or collagen based vascular closure device placement within 90 days of procedure.
   * No prior femoral artery needle puncture within 30 days of procedure.
   * No current active localized groin infection, traumatic vascular injury, femoral artery aneurysm, arteriovenous (AV( fistula, or pseudoaneurysm.
8. Patient must be willing to comply with all required follow-up exams.

Exclusion Criteria:

1. Patient has a need for emergent surgery.
2. Patient has a dissecting aneurysm.
3. Patient has an acutely ruptured aneurysm.
4. Patient has an acute vascular injury.
5. Patient has had a previous repair of the abdominal aortic aneurysm or the iliac artery.
6. Patient has a mycotic aneurysm or has an active systemic infection.
7. Patient has unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina, or onset of prolonged angina).
8. Patient has unstable peripheral artery disease with critical limb ischemia (CLI).
9. Patient has congestive heart failure (CHF). Subjects in Class I or II will be allowed to participate in the protocol, subjects in Class III or IV should be excluded. The New York Heart Association NYHA Functional Classification is used as a reference, see Appendix III.
10. Patient has had a myocardial infarction (MI) and/or stroke (CVA) within the past 3 months.
11. Patient requires use of techniques (e.g. Chimney graft) that would cover the renal arteries.
12. Patient requires planned adjunctive devices (e.g. renal stents) to complete the procedure.
13. Patient has a major surgical or interventional procedure planned during or within ± 30 days of the AAA repair.
14. Patient has history of connective tissue disease (e.g., Marfan's or Ehler's-Danlos syndrome).
15. Patient has history of bleeding disorders or refuses blood transfusions.
16. Patient has dialysis dependent renal failure or baseline serum creatinine level >2.0mg/dl.
17. Patient has a known hypersensitivity or contraindication to anticoagulation or contrast media that is not amenable to pre-treatment.
18. Patient has a known allergy or intolerance to polytetrafluoroethylene (PTFE), PEG- based polymers, fluorinated ethylene propylene (FEP) or nitinol.
19. Patient is on home oxygen.
20. Patient is morbidly obese (BMI ≥ 40 kg/m2).
21. Patient was admitted from a skilled nursing facility.
22. Patient has a limited life expectancy of less than 1 year.
23. Patient has an inability to be discharged within 1 day (one midnight stay) of the procedure. Examples included but are not limited to, comorbid conditions, unable to admit the day of procedure, live too far away from treatment center, or insufficient post-operative family support.
24. Patient is currently participating in an investigational device or drug clinical trial.
25. Patient has other medical social or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll male and female subjects 18 years of age and older that have an AAA and meet all other inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Major Adverse Events | 30 days

SECONDARY OUTCOMES:
Serious and Non-Serious Adverse Events, including vascular and major access site vascular complications | 30 days
Access Technical Success, defined as percent of procedures successfully completed with bilateral percutaneous access | 30 days
Treatment Success, defined as percent of subjects who successfully follow least invasive protocol through discharge | 30 days
Blood loss, including if transfusion required | 30 days
Percent of procedures completed without general anesthesia | 30 days
Anesthesia Time | 30 days
Procedure Time | 30 days
Contrast Volume | 30 days
Fluoroscopy Time | 30 days
Time to hemostasis | 30 days
Time to ambulation | 30 days
Time to normal diet | 30 days
Groin pain via Wong-Baker FACES Pain Rating Scale- a 10-point visual analog scale (0=none; 10= worst imaginable) | 30 days
Quality of Life via the EuroQol Group's EQ-5D form | 30 days
Percent of subjects discharged without ICU admission | 30 days
Length of ICU Stay, if required | 30 days
Length of hospital stay | 30 days
Percent of subjects discharged within only one midnight stay | 30 days
Freedom from Type I and III endoleaks | 30 days
Freedom from AAA rupture | 30 days
Freedom from conversion to open repair | 30 days
Freedom from AAA related secondary interventions | 30 days
Freedom from mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Randolph P. Guzman, MD, Principal Investigator — St. Boniface Hospital
Locations (1):
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada